CLINICAL TRIAL: NCT01297842
Title: An Open-label, Randomized Equivalence Trial and Cost-effectiveness Analysis of Ertapenem Versus Other Carbapenems for Treatment of Extended -Spectrum Beta-Lactamase (ESBL)-Producing Gram-negative Bacterial Infections
Brief Title: Ertapenem Versus Meropenem/Imipenem for ESBL+ Gram-negative Infections
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Visanu Thamlikitkul, Division of Infectious Diseases and tropical medicine, Department of medicine, Faculty of Medicine Siriraj Hospital., Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SirirajCEU 54-001
Record Dates: First submitted 2011-02-14; First posted 2011-02-17 (Estimated); Last update posted 2012-01-02 (Estimated); Status verified 2011-12

CONDITIONS: Drug Safety
MeSH Terms: interventions — Ertapenem; Meropenem; Imipenem; Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ertapenem (Experimental): Ertapenem 1 gram per day for 7 to 14 days
  Interventions: Drug: Ertapenem
- Meropenem or Imipenem (Active Comparator): Meropenem or Imipenem o.5 or 1 gram 3 to 4 times a day for 7 to 14 days
  Interventions: Drug: Meropenem or Imipenem

INTERVENTIONS:
Drug: Ertapenem — Ertapenem 1 gram per day for 7 to 14 days
  Other Names: Invanz
  Arms: Ertapenem
Drug: Meropenem or Imipenem — Meropenem or Imipenem 0.5 to 1 gram 3 to 4 times per day for 7 to 14 days
  Other Names: Meronem; Tienam
  Arms: Meropenem or Imipenem

SUMMARY:
Adult patients with ESBL-producing Gram negative infections are randomized to receive ertapenem or meropenem/imipenem. Clinical and microbiological responses between both groups are compared.

DETAILED DESCRIPTION:
Ertapenem is active against ESBL-producing Gram negative bacteria. This study is conducted to determine if ertapenem is effective against ESBL-producing Gram negative infections similar to meropenem/imipenem.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients aged >18 years with documented ESBL +ve GNB infection
* Receive meropenem or imipenem/cilastatin as empiric antibiotic therapy

Exclusion Criteria:

* Having been treated with meropenem or imipenem/cilastatin for longer than 72 hours
* Have active P. aeruginosa co-infection
* Pregnancy or breast feeding
* Allergy to carbapenems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-04 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with cure or improvement | 14 days
  Cure Improvement Persistence Death from Infection

SECONDARY OUTCOMES:
Number of subjects with eradication of the causative bacteria | 14 days
  Eradication Persistence Superinfection

CONTACTS AND LOCATIONS:
Overall Officials: Visanu Thamlikitkul, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Rattanaumpawan P, Werarak P, Jitmuang A, Kiratisin P, Thamlikitkul V. Efficacy and safety of de-escalation therapy to ertapenem for treatment of infections caused by extended-spectrum-beta-lactamase-producing Enterobacteriaceae: an open-label randomized controlled trial. BMC Infect Dis. 2017 Mar 1;17(1):183. doi: 10.1186/s12879-017-2284-1. PMID 28249572